CLINICAL TRIAL: NCT07013760
Title: Observational Retrospective Study to Characterize and Assess Clinical Outcomes of Patients Receiving Tezepelumab After Marketing Approval in Spain
Brief Title: Characterize and Assess Clinical Outcomes of Patients Receiving Tezepelumab After Marketing Approval in Spain
Acronym: T-ROSS-II
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00038
Record Dates: First submitted 2025-04-04; First posted 2025-06-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational retrospective study to characterize and assess clinical outcomes of patients receiving tezepelumab after marketing approval in Spain

DETAILED DESCRIPTION:
T-ROSS-II has been designed to conduct a new observational study to generate additional evidence on the use of tezepelumab in severe asthma patients in routine clinical practice in Spain after its launch.

This is an observational, multi-centre, retrospective, single-arm study in patients 12 years and older with severe asthma.

Approximately 400 patients meeting the study eligibility criteria will be included in the T-ROSS-II.

ELIGIBILITY:
Inclusion Criteria:

Patients who received at least 1 tezepelumab dose after commercialization in Spain diagnosed with severe asthma who are inadequately controlled with high-dose inhaled corticosteroids and a long-acting β2-agonist ± additional medications for asthma control.

* Patients aged ≥12 years at the index date.
* Patients with continuous enrolment in the data source for at least 12-months before the index date.
* Patients with at least three months of continuous enrolment in the data source after the index date.

Exclusion Criteria:

Patients who received tezepelumab or any biologic drug for the treatment of asthma in a clinical trial at any time during the 12-months prior to the index date*.

• Patients who had initiated 3 or more non-tezepelumab biologic treatment (omalizumab, mepolizumab, reslizumab, benralizumab and dupilumab) for severe asthma at any time prior to the index date).

Ages: 12 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of all the patients ≥ 12 years old who have received tezepelumab according to the usual clinical practice under the discretion of the physician according with the European SmPc and the reimbursement conditions in Spain between October 1st 2023 and 12 months before the site initiation, who meet all the inclusion criteria and none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Socio-demographic variables: Age (years), Gender (male, female, other); Smoking status (Current smoker, Ex- smoker, Non-smoker) and cumulative index (packs/year); Height (cm) and weight (kg); Body Mass Index (BMI) (kg/m 2 ) | Index date (treatment initiation with tezepelumab)
  To describe the demographic characteristics of patients
Exacerbation (number of exacerbations) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
Comorbidities (e.g., allergic rhinitis, nasal polyposis, gastroesophageal reflux, chronic obstructive pulmonary disease (COPD), atopic dermatitis and other eosinophilic conditions, conditions related to OCS chronic use, etc.) | From 12 months before index date until index date (defined as the date of treatment initiation with tezepelumab)
Number of respiratory infections and diseases in the previous 12 months and index date | From 12 months before index date until index date (defined as the date of treatment initiation with tezepelumab)
Number of participants with an Allergy test (Prick test, RAST or similar, clinical relevance of allergy, etc.) (only baseline) | Only on the baseline (12 months prior to Index date)

SECONDARY OUTCOMES:
Asthma Control Test (ACT) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  A short, simple, patient-based tool for identifying subjects with poorly controlled asthma. ACT assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. The seores range from 5 (poor control of asthma) to 25 (complete control of osthmo), with higher seores reflecting greater asthma control. An ACT score >19 indicates well controlled asthma. The investigators will use the Spanish validation
Lung function measurements | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  Lung function measurements including spirometry (FEV1 (L))
FeNO (ppb) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
Blood neutrophil count (109 /L, mm^3) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
IgE (IU/mL) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
Asthma Impairment and Risk Questionnaire (AIRQ) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  The score range from 1 to 10. Scores from 0-1 indicate well controlled-asthma. From 2-4 no well-controlled and ≥ 5 bad control.
Asthma Quality of Life Questionnaire (AQLQ) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  It is a validated scale with 32 questions. The questions are scored on a scale of 1- 7, with higher scores indicating better quality of life.
MiniAQLQ (Mini Asthma Quality of Life Questionnaire) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  This instrument has 15 questions. The questions are scored on a scale of 1- 7, with higher scores indicating better quality of life.
SNOT-22 (Sino-Nasal Outcome Test) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)
  It consists of 22 items, rated from 0 ('no problem at all') to 5 ('worst possible symptom'). Possible SNOT-22 total-scores range from 0 to 110, with higher SNOT-22 total-scores indicating worse symptoms.
Blood eosinophil count (BEC) (109 /L, mm^3) | From 12 months before index date (defined as the date of treatment initiation with tezepelumab) until the end of the follow up which will start after index date and will last up to inclusion (the period will last 9-15 months depending on inclusion date)

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Research Site, Andalucia
  - Research Site, C. Valenciana
  - Research Site, C. Y Leon
  - Research Site, Cantabria
  - Research Site, Castilla La Mancha
  - Research Site, Cataluna
  - Research Site, Extremadura
  - Research Site, Galicia
  - Research Site, Islas Canarias
  - Research Site, Madrid
  - Research Site, Navarra
  - Research Site, Pais Vasco

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/